CLINICAL TRIAL: NCT06521450
Title: Concurrent Surgery for Prolapse Repair and Stress Urinary Incontinence to Reduce the Risk of Postoperative Surgical Intervention for Incontinence
Brief Title: Concurrent Surgery for Prolapse and Stress Urinary Incontinence to Reduce Further Surgery for Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sheema Yousuf, Doctor, Shalamar Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-693-4
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- combined surgery group (Active Comparator)
  Interventions: Procedure: anti incontinence surgery
- prolapse surgery only group (Active Comparator)
  Interventions: Procedure: anti incontinence surgery

INTERVENTIONS:
Procedure: anti incontinence surgery — anti incontinence surgery with prolapse surgery will be performed simultaneously

SUMMARY:
Urinary incontinence is a common and distressing medical condition which affects 26% of women in developing countries.Globally upto 54% women suffer from pelvic organ prolapse and stress urinary incontinence concomitantly.Women with coexisting stress incontinence have a 40% risk of undergoing subsequent surgery for postoperative stress incontinence and woem with occult incontinence have a 15% risk.Overall,there is sufficient evidence that for women who are symptomatic of stress incontinence and prolapse,concomitant vaginal surgery for both problems is beneficial for reducing postoperative incontinence.However,it must be borne in mind that in woen undergoing vaginal prolapse surgery alone,almost 1/3 may experience cure of incontinence symptoms and despite concomitant continence surgery,stress urinary incontinence persist in approximately 1/3 of women.This study will be conducted to assess whether women with polpase and stress urinary incontinence could benefit from combined surgery in regards of requiring further surgery for stress incontinence.

DETAILED DESCRIPTION:
INTRODUCTION

Urinary incontinence (UI), is a common and distressing medical condition which affects 26% of women in developing countries and stress urinary incontinence (SUI) (12.6%) is the most common type.1 One of the important risk factors for SUI is pelvic organ prolapse.2 Pelvic organ prolapse(POP) is descent of pelvic organs resulting in protrusion of pelvic structures including bladder, rectum and uterus beyond their anatomical confines. In low and middle-income countries, the prevalence of pelvic organ prolapse is 19.7% (estimated range is 3.4%-56.4%).3 In a study, the prevalence of prolapse in Pakistan was 10.3%.4 Globally in up to 54 % of women, pelvic organ prolapse and stress incontinence coexists.5 In Pakistan 12.5% women will suffer with both prolapse and urinary incontinence.2

Patients showing no improvement with conservative measures are offered surgery. The surgical methods used for SUI include Burch colposuspension (BC), tension-free vaginal tape (TVT)and trans obturator tape (TOT).6 For prolapse the route of repair can be abdominal or vaginal and surgical methods include reconstructive procedures preserving uterus or vaginal hysterectomy.7 The uterus preserving surgeries include Sacrohysteropexy (ASC), sacrospinous ligament fixation, ventrosuspension and Manchester repair.8,9

Many women undergoing surgery for pelvic organ prolapse (POP) will experience incontinence after prolapse repair. Developing incontinence after prolapse repair is even more common among women with urinary incontinence before the surgery.10 In a recent study women with coexisting SUI have a 40% risk of undergoing subsequent surgery for postoperative SUI and women with occult SUI have a 15% risk. 10 It is shown in some studies that women could have lower risk of subsequent continence surgery for SUI after combination surgery than after prolapse surgery only.11 However, another study showed that about a third of women with POP and SUI will experience resolution of SUI symptoms following isolated POP repair.12,13 Van der Ploeg et al. conducted a large multicentre RCT, and results showed a significant reduction in postoperative SUI rates in the combined surgery group as compared to POP repair only; 22% versus 61% .Despite 61% of women reporting postoperative SUI in the POP repair-only group, only 17% went on to receive surgical treatment for SUI within 12 months of follow-up. Potential explanations include the use of alternative non-surgical treatments, the SUI not being severe enough to warrant surgery, or the woman's desire to avoid further surgery and operative risks. 14 Costantini et al. evaluated concomitant colposuspension at the time of abdominal sacrocolpopexy surgery versus sacrocolpopexy alone and showed no significant benefit in adding Burch colposuspension.15 Overall, there is sufficient evidence that for women who are symptomatic of SUI and POP, concomitant vaginal POP repair and anti-incontinence surgery is beneficial for reducing postoperative SUI. However, it must be borne in mind that in women undergoing vaginal POP surgery alone, almost one-third may experience cure of SUI symptoms and despite concomitant continence surgery, SUI can still persist in approximately one-third of women.16 So, we aim to compare the risk of surgical intervention for stress urinary incontinence after combined prolapse and anti-incontinence surgery and prolapse surgery alone.

RATIONALE:

Urinary incontinence (UI), is a common and distressing medical condition which affects 26% of women in developing countries.1Globally in up to 54 % of women pelvic organ prolapse and stress incontinence coexists.2 Women with coexisting SUI have a 40% risk of undergoing subsequent surgery for postoperative SUI and women with occult SUI have a 15% risk. Overall, there is sufficient evidence that for women who are symptomatic of SUI and POP, concomitant vaginal POP repair and anti-incontinence surgery is beneficial for reducing postoperative SUI. However, it must be borne in mind that in women undergoing vaginal POP surgery alone, almost one-third may experience cure of SUI symptoms and despite concomitant continence surgery, SUI can still persist in approximately one-third of women.16

OBJECTIVE:

This study will assess whether women with POP and stress urinary incontinence could benefit from combined surgery in regards of requiring further surgery for SUI.

OPERATIONAL DEFINITIONS Stress Urinary Incontinence(SUI): Involuntary leakage of urine when there is raised intraabdominal pressure such as during coughing, weight lifting etc.1 Pelvic organ prolapse (POP): Uterine prolapse occurs when pelvic floor muscles and ligaments stretch and weaken until they no longer provide enough support for the uterus resulting in protrusion of pelvic organs beyond their anatomical position.2,6 Pelvic organ prolapse quantification system (POP-Q): It is used to subjectively quantify the stage of prolapse.6 Paralytic ileus: It is a condition in which there is a functional motor paralysis of the digestive tract secondary to neuromuscular failure resulting in abdominal distension, absent bowel sounds and electrolyte imbalance.6 Urinary retention: Inability to pass urine despite persistent effort resulting in painful and palpable bladder or chronic high post void residual urine >300ml as defined by international continence society.

Dysuria: Sensation of pain, burning stinging or itching of the urethra associated with urination.2,3,4 Wound infection: It is the presence of replicating microorganisms within a wound leading to tissue injury resulting in either purulent discharge, pain, tenderness, localised swelling or redness.2,3,4 Blood loss >500ml: Blood loss will be quantified by using gravimetric method which is measuring irrigation fluid and weighing surgical sponges and subtracting the dry weight to obtain a blood volume measurement.17

MATERIAL AND METHODS Settings: Department of Urogynaecology Shalamar Hospital, Lahore Study design: Randomized controlled trial Study Population: Adult females 41-83 years age presenting with pelvic organ prolapse and stress urinary incontinence.

Duration of study: The duration of study will be six months after ethical approval.

Sampling Technique: Simple random sampling

Sample size Calculation/Statistical power:

n=Z2 x p x (1-p)÷E2 n is sample size Z is Z value (the number of standard deviation from the mean) for the desired confidence level (for 95%, Z is 1.96) P is the estimated proportion of the population that has the characteristic of interest (in this case 40% or 0.40) E is the margin of error (5% or 0.05) p =0.40 E =0.05 Z =1.96 n =1.962 x 0.40 x (1-0.40)/0.052 1.962 =3.8416

First, we calculate the numerator:

0.40x (1-0.40) =0.40x0.60=0.24 Now, multiply these together 3.8416x0.24=0.921984

Next, we calculate the denominator:

0.052=0.0025

Finally, we divide the numerator by the denominator to get the sample size:

n =0.921984/0.0025 = 368.7936 n/ = n ÷1+n-1 /N where n/ is the adjusted sample size for the finite population n is the initial sample size calculated using the formula for an infinite population N is the total population size

Given:

n=369(initial sample size) N=200(total population size) n/ = 369 ÷1+369-1 /200 n/ =369/2.84=129.93 since the sample size must be a whole number, we round up to the nearest whole number: n/ =130

Inclusion Criteria: Adult females 41-83 years age presenting with concurrent prolapse and stress urinary incontinence willing to participate in the study.

Exclusion criteria: Study exclusion criteria will be urge incontinence according to questionnaire, urinary tract infection, unwilling for surgery, unfit for surgery, urogenital malignancy, urolithiasis.

Procedure/methods in detail:

A total of 130 patients between ages of 41 and 83 years fulfilling the selection criteria will be included in the study. It will be a randomised controlled study of prolapse surgery with or without anti-incontinence surgery. Patients presenting with stress urinary incontinence and prolapse will be enrolled in the study. Patients will be randomly assigned to either combined surgery group or POP alone group, each group will have 65 patients. All patients will give written informed consent for study participation, and approval for the study will be obtained from the ethical committee of our hospital. All women will undergo preoperative assessments involving detailed medical and surgical histories. Baseline characteristics will be recorded on specially designed proforma. Participation in the study will be voluntary and all patients will have free choice to withdraw from the study at any stage which will not affect their management. In all patients SUI will be visualized after performing physical examination with cough stress test and prolapse will be staged by using pelvic organ prolapse quantification system(POP-Q). A cough stress test will be performed in the supine position with the bladder comfortably filled with about 250mL of urine. Severity of stress urinary incontinence will be assessed by a severity index score. Severity index will be created by multiplying the reported frequency (four levels) by the amount of leakage (two levels) (annexure I). The resulting index value (1-8) will be further categorised into slight (1-2), moderate (3-4), and severe (6-8).18

The operation will be performed under spinal or general anaesthesia, according to patients and surgeon preference. The same surgeon will perform all the surgeries. Cystoscopy will be performed for all patients at the end of procedure to identify any bladder injury. Any intra-operative complications like blood loss > 500 ml and visceral injury (ureter, bowel, bladder) will be noted and managed accordingly. Routine post-operative care will be provided and any complications like paralytic ileus, urinary retention, dysuria and wound infection will be noted and treated.

The primary outcome will be symptomatic stress urinary incontinence (SUI) requiring continence surgery at 6 months. Secondary outcome measures will be quality of life parameters. Quality of life (QOL) will be assessed with the International Consultation on Incontinence Questionnaire short form (ICIQ-UI SF). The questionnaire will be filled before and after surgery for all patients. Total score range will be 0-21(slight 1-5, moderate 6-12, severe 13-18, very severe 19-21). They will be examined and questioned about their satisfaction with the surgery at each follow up visit. Patient follow-up will take place at 1 week, 6 weeks and 6 months. In the visits 1 week and 6 weeks after surgery, wound healing will be checked. In the visit 6 months after surgery, a cough stress test will be performed for objective assessment. Objective cure will be defined as a negative cough stress test. 'Failure'' will be defined as a positive cough stress test.

Data analysis:

All data will be analysed using SPSS version 21. Continuous variables including age, BMI, parity, duration of surgery, blood loss during surgery and days of hospital stay will be presented as mean ± SD. Categorical variables including prolapse stage, complications (injury to ureter, bowel, bladder, paralytic ileus, urinary retention, dysuria, wound infection) and patient's satisfaction with the results of procedure will be presented as frequencies and percentages. Pre-and postoperative questionnaire data will be analysed with Student's t test. A p value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult females 41-83 years age presenting with concurrent prolapse and stress urinary incontinence willing to participate in the study.

Exclusion Criteria:

- Exclusion criteria: Study exclusion criteria will be urge incontinence according to questionnaire, urinary tract infection, unwilling for surgery, unfit for surgery, urogenital malignancy, urolithiasis.

Ages: 41 Years to 83 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
symptomatic stress urinary incontinence requiring surgery at six months | at six months after surgery

SECONDARY OUTCOMES:
quality of life parameters.It will be assessed using ICIQ-UI short form questionnaires | 1 week,6 week and six month after surgery
  0-12 score will show improved quality of life while 13-21 will show impaired quality

IPD SHARING:
Plan to Share IPD: No